CLINICAL TRIAL: NCT02765087
Title: Diagnostic Utility of the E-Nose for Pleural TB
Brief Title: E-Nose: Diagnostic Tool for Pleural TB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Central de Venezuela (Other)
Collaborators: The ENose Company, Zutphen, Netherlands (Unknown); Foundation for Research in Mycobacteria (FUNDAIM) (Other)
Responsible Party: Principal Investigator, Jacobus H. de Waard, Chief of Tuberculosis Laboratory, Universidad Central de Venezuela
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EN002
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Tuberculosis, Pleural
MeSH Terms: conditions — Tuberculosis, Pleural | interventions — Health Records, Personal; Electronic Nose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pleural TB (Experimental): This group consist of patients with TB pleural effusion.
  Intervention:
  1. Inform Consent
  2. Medical History
  3. E-Nose Device
  4. Chest CT
  5. Cytomorphologic & Cytochemistry of pleural Fluid.
  6. Adenosine Deaminase value of pleural Fluid.
  Interventions: Other: Medical History; Device: E-Nose; Other: Chest CT; Other: Pleural Fluid Analysis
- Control (Active Comparator): Patients with pleural effusion with different aetiologies than Tuberculosis.
  Intervention:
  1. Inform Consent
  2. Medical History
  3. E-Nose Device
  4. Chest CT
  5. Cytomorphologic & Cytochemistry of pleural Fluid.
  6. Adenosine Deaminase value of pleural Fluid.
  Interventions: Other: Medical History; Device: E-Nose; Other: Chest CT; Other: Pleural Fluid Analysis

INTERVENTIONS:
Other: Medical History — Oriented Survey and complete physical exam.
Device: E-Nose — Patient will breath trough the device for 5 minutes, and during and after the intervention will be assessed for adverse effects related to the use of the e-Nose, according to the CTCEA
Other: Chest CT
Other: Pleural Fluid Analysis — Cytomorphology Cytochemistry Adenosine Deaminase Value

SUMMARY:
The purpose of this study is to determine the diagnostic utility of the device 'Electronic Nose' for Pleural TB, which is a Extra pulmonary TB form, compared with pleural biopsy, the current gold standard.

DETAILED DESCRIPTION:
The aim of the study is to determine the diagnostic utility of the device 'Electronic Nose' for Pleural TB, which is a Extra pulmonary TB form.

The patient who qualified for the study, according to the inclusion criteria, after consenting, will be guided through and oriented survey for risk factors, then a complete physical exam, and after that, the patient will breathe for 5 minutes trough the device, which stores the patient information, that later will be download to a computer and will be send to the server's manufacturer company, in Netherlands.

During and after the use of the device, investigators determine the adverse effects of the intervention, according to the CTCEA.

Investigators use the pleural biopsy, which is the gold standard, to determine the diagnostic utility of the test. And, will compare the results with other tests currently perform as the regular diagnostic routine, such as Chest CT, adenosine deaminase value of pleural fluid and cytomorphologic & cytochemistry of the pleural fluid.

Patient Registries will be keep in an electronic database, as well as handwriting history, with the backup copy in the records of the hospital in which the patient was admitted.

Auditories will be realised by the Ethics Committee in different time frames.

ELIGIBILITY:
Inclusion Criteria

1. Accept to participate in the study through a signed informed consent approved by the Ethical Committee of our Institution.
2. More than 15 years old.
3. Pleural effusion of any etiology

Exclusion Criteria:

1. Severe compromise of the general condition
2. Not capable to exhaled through the E-nose.
3. No possibility to follow-up.
4. By discretion of the research team.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the device for the diagnosis of Tuberculosis Pleural effusion | 1 year

SECONDARY OUTCOMES:
Adverse Effects related to the use of the device, according to the CTCEA | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacobuss de Waard, PhD., Principal Investigator — Instituto de Biomedicina
Locations (1):
- Instituto de Biomedicina, Caracas, DC, Venezuela

IPD SHARING:
Plan to Share IPD: No